CLINICAL TRIAL: NCT02106455
Title: Sodium Risedronate 17.5 mg Tablets Special Drug Use Surveillance in Patients With Osseous Paget's Disease (All-case Surveillance) - 48-week Surveillance -
Brief Title: Sodium Risedronate Tablets - Special Drug Use Surveillance in Patients With Osseous Paget's Disease (All-case Surveillance) -48-week Surveillance -
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 067-211; JapicCTI-142480 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Osseous Paget's Disease
Keywords: Pharmacological theapy
MeSH Terms: conditions — Osteitis Deformans | interventions — Risedronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 17.5 mg of sodium risedronate: 17.5 mg of sodium risedronate is administered orally with a sufficient volume (approximately 180 mL) of water once daily after waking for 8 consecutive weeks.
  Interventions: Drug: Sodium risedronate

INTERVENTIONS:
Drug: Sodium risedronate — Sodium risedronate tablets
  Other Names: Benet 17.5mg Tablets; Actonel 17.5mg Tablets

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of sodium risedronate tablets administered once daily (one tablet per dose) in patients with osseous Paget's disease for 48 weeks from baseline in daily medical practice.

DETAILED DESCRIPTION:
This special drug use surveillance was designed to evaluate the safety and efficacy of sodium risedronate tablets 17.5 mg administered once daily (one tablet per dose) in patients with osseous Paget's disease in daily medical practice.

The usual dosage for adults is 17.5 mg of sodium risedronate administered orally with a sufficient volume (approximately 180 mL) of water once daily after waking for 8 consecutive weeks. For at least 30 minutes after administration, participants should avoid lying in a supine position and taking food, drink (except for water) or other oral drugs.

ELIGIBILITY:
Inclusion Criteria:

* Osseous Paget's disease patients treated with sodium risedronate tablets 17.5 mg

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Osseous Paget's disease
Sampling Method: Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 92 investigative sites in Japan, from 01 August 2008 to 24 October 2017.
Pre-assignment Details: Participants with a historical diagnosis of osseous Paget's disease were enrolled. Participants received interventions as part of routine medical care.
Groups:
- Sodium Risedronate 17.5 mg: 17.5 mg of sodium risedronate was administered orally with a sufficient volume (approximately 180 mL) of water once daily after waking for 8 consecutive weeks. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Sodium Risedronate 17.5 mg
Started | 315
Completed | 307
Not Completed | 8
Not completed — Case Report Form Uncollected | 6
Not completed — Protocol Deviation | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 304
    (all) | 63.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134
  Male | 173
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 307
Pregnancy Status (not pregnant) [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    number analyzed (Participants) | 134
    (all) | 134
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 167
    (all) | 159.49 (9.78)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 170
    (all) | 59.74 (12.04)
Classification by Treatment History [Count of Participants; unit: Participants]
  Initial Treatment | 184
  Repetitive Treatment | 123
Treatment Duration [Count of Participants; unit: Participants]
  ≤ 56 Days | 145
  ≥ 57 Days | 159
  Unknown | 3
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient, inpatient, and outpatient and inpatient.
  Participants
    Outpatient | 288
    Outpatient and Inpatient | 19
Detailed Diagnosis of Osseous Paget's Disease [Count of Participants; unit: Participants]
  Monostotic Osseous Paget's Disease | 125
  Polyostotic Osseous Paget's Disease | 176
  Undifferentiated/Unknown | 6
Duration of Diagnosis of Osseous Paget's Disease [Count of Participants; unit: Participants] — Mean duration between start of study and first time of diagnosis of Osseous Paget's Disease was reported.
  Participants
    < 1 Year | 106
    1 to < 5 Years | 60
    ≥ 5 Years | 71
    Unknown (Not Reported) | 70
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Presence of Medical Complications | 105
    Had Presence of Medical Complications | 202
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had No Medical History | 156
    Had Medical History | 150
    Unknown | 1
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had No Predisposition to Hypersensitivity | 290
    Had Predisposition to Hypersensitivity | 9
    Unknown | 8
Family History of Osseous Paget's Disease [Count of Participants; unit: Participants] — Reported data were the numbers of participants who had/did not have family with historical diagnosis of osseous Paget's disease.
  Participants
    Had No Family History | 231
    Had Family History | 7
    Unknown | 69
Experience of Fracture at Disease Site [Count of Participants; unit: Participants] — Reported data were the numbers of participants who had/did not have experience of fracture at disease site of osseous Paget's disease.
  Participants
    Had No Experiences | 274
    Had Experience | 33
Past Drug Therapy for Osseous Paget's Disease [Count of Participants; unit: Participants] — Reported data were the numbers of participants who had/did not have received drug therapies for osseous Paget's disease in the past before the start of this study.
  Participants
    Had No Therapies | 92
    Had Therapy | 209
    Unknown | 6
Concurrent Medication [Count of Participants; unit: Participants]
  Had No Concurrent Medication | 134
  Had Concurrent Medication | 173

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Drug Reactions
Description: Adverse drug reaction refers to adverse events related to administered drug.
Time Frame: Up to 48 weeks
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 307
Percentage of Participants | 14.98

2. Secondary Outcome: Percentage of Changes From Baseline in Excess Serum Alkaline Phosphatase (ALP) Level at Final Assessment Point
Description: Percentage of changes from baseline in excess serum ALP level at final assessment point (up to 48 weeks) was reported.
Time Frame: Baseline and final assessment point (Up to 48 weeks)
Population: Efficacy assessment population; The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. The number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 251
Percentage of change | -72.47 (125.78)

3. Secondary Outcome: Percentage of Changes From Baseline in Serum ALP Level at Final Assessment Point
Description: Percentage of changes from baseline in serum ALP level at final assessment point (up to 48 weeks) was reported.
Time Frame: Baseline and final assessment point (Up to 48 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 251
Percentage of change | -31.71 (30.47)

4. Secondary Outcome: Number of Participants Stratified by Comparison of Pain Scale Associated With Osseous Paget's Disease Between Baseline and Final Assessment Point
Description: Investigators marked severity of pain with a 4-point scale ranging from "None" to "Very Severe" (None, Mild, Severe, Very Severe) at baseline and the final assessment point. This scale was specified on the protocol of this observational study. The reported data were number of participants stratified by comparison of pain severity between baseline and final assessment point described as "None (at baseline) to Severe (at final assessment point)".
Time Frame: Baseline and final assessment point (Up to 48 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 258
Participants
  None to None | 138
  None to Mild | 1
  None to Severe | 1
  Mild to None | 12
  Mild to Mild | 14
  Severe to None | 18
  Severe to Mild | 21
  Severe to Severe | 39
  Severe to Very Severe | 1
  Very Severe to None | 6
  Very Severe to Mild | 2
  Very Severe to Severe | 4
  Very Severe to Very Severe | 1

5. Secondary Outcome: Number of Participants Stratified by Assessment of Image Findings of Bone Morphogenic Abnormalities at Final Assessment Point Compared With Baseline
Description: Investigator marked assessment of image findings of bone morphogenic abnormalities at final assessment point compared with baseline as follows; "improved", "unchanged", "worsened". The reported data were the number of participants stratified by assessment of image findings at final assessment point.
Time Frame: Baseline and final assessment point (Up to 48 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 74
Participants
  Improved | 7
  Unchanged | 66
  Worsened | 1

6. Secondary Outcome: Number of Participants Stratified by Assessment of Image Findings of Trabecular Bone Structural Abnormalities at Final Assessment Point Compared With Baseline
Description: Investigator marked assessment of image findings of trabecular bone structural abnormalities at final assessment point compared with baseline as follows; "improved", "unchanged", "worsened". The reported data were the number of participants stratified by assessment of image findings at final assessment point.
Time Frame: Baseline and final assessment point (Up to 48 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 72
Participants
  Improved | 14
  Unchanged | 57
  Worsened | 1

7. Secondary Outcome: Number of Participants Stratified by Assessment of Image Findings of Other Abnormalities at Final Assessment Point Compared With Baseline
Description: Other Abnormalities refer to bone abnormal findings excluding bone morphogenic abnormalities and trabecular bone structural abnormalities (see Outcome Measure 5 and 6). Investigator marked assessment of image findings of other abnormalities at final assessment point compared with baseline as follows; "improved", "unchanged", "worsened". The reported data were the number of participants stratified by assessment of image findings at final assessment point.
Time Frame: Baseline and final assessment point (Up to 48 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 39
Participants
  Improved | 6
  Unchanged | 31
  Worsened | 2

8. Secondary Outcome: Percentage of Changes From Baseline in Urinary Type 1 Collagen Cross-Linked N-telopeptide (Urinary NTX) Level at Final Assessment Point
Description: Percentage of changes from baseline in urinary NTX level at final assessment point (up to 48 weeks) was reported. Urinary NTX is one of bone metabolism markers.
Time Frame: Baseline and final assessment point (Up to 48 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 42
Percentage of change | -51.01 (34.43)

9. Secondary Outcome: Percentage of Changes From Baseline in Urinary Deoxypyridinoline (Urinary DPD) Level at Final Assessment Point
Description: Percentage of changes from baseline in urinary DPD level at final assessment point (up to 48 weeks) was reported. Urinary DPD is one of bone metabolism markers.
Time Frame: Baseline and final assessment point (Up to 48 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 30
Percentage of change | -10.01 (60.23)

10. Secondary Outcome: Percentage of Changes From Baseline in Serum Bone Alkaline Phosphatase (Serum BAP) Level at Final Assessment Point
Description: Percentage of changes from baseline in serum BAP level at final assessment point (up to 48 weeks) was reported. Serum BAP is one of bone metabolism markers.
Time Frame: Baseline and final assessment point (Up to 48 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 52
Percentage of change | -43.57 (33.13)

11. Secondary Outcome: Percentage of Participants Stratified by Treatment Compliance (Medicine Adherence) During Treatment Period
Description: Treatment compliance of this outcome measure refers to the percentage of participants who correctly follow medication. The reported data are percentage of participants in the classification including 4 specific degrees of treatment compliance; 90 % or more; 67 % or more and <90 %; 25 % or more and <67 %; less than 25 % or "unknown".
Time Frame: Up to 48 weeks
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Sodium Risedronate 17.5 mg
Number analyzed (Participants) | 307
Percentage of participants
  90 % or More | 95.11
  67 % or More and <90 % | 2.61
  25 % or More and <67 % | 0.65
  Less than 25 % | 0.33
  Unknown | 1.30

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Description: Only adverse drug reactions (ADRs) were collected in this study. ADRs are adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms/diseases temporally associated with the use of a medicinal product reported throughout the study.
Arm/Group | Sodium Risedronate 17.5 mg
All-Cause Mortality (participants affected / at risk) | 0/307
Serious Adverse Events (participants affected / at risk) | 15/307
Other Adverse Events (participants affected / at risk) | 14/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Risedronate 17.5 mg (N=307)
Pneumonia (Infections and infestations) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Cerebral infarction (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Risedronate 17.5 mg (N=307)
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT02106455/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT02106455/SAP_001.pdf